CLINICAL TRIAL: NCT01633541
Title: Concomitant Chemotherapy AND Bcl-xL Inhibitor (AT-101) For Bio-selection For Organ Preservation In Patients With Advanced Laryngeal Cancer
Brief Title: Chemotherapy AND Bcl-xL Inhibitor (AT-101) For Organ Preservation In Adults With Advanced Laryngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2010.101; HUM00043975 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Laryngeal Cancer
MeSH Terms: conditions — Laryngeal Neoplasms | interventions — gossypol acetic acid; Docetaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- platinum/docetaxel + AT-101 (Experimental): platinum/docetaxel + AT-101 The platinum will either be cisplatin or carboplatin as deemed best by the medical oncologist.
  (Both Arms) Day #1: Patients will undergo induction chemotherapy with (TP) docetaxel (Taxotere) 75 mg/m2 and cisplatin 100 mg/m2 (or Carboplatin AUC 6).
  (AT-101 Arm) Days #1-3: Patients will receive AT-101 40 mg orally twice daily On Day 23 (+/- 3 days), there will be a direct laryngoscopy (DL) with tumor biopsy and blood draw, repeat CT scan of the neck with perfusion within a week biopsy.
  Interventions: Drug: AT-101; Drug: Cisplatin; Drug: Carboplatin
- Active Comparator arm (Active Comparator): (Both Arms) Day #1: Patients will undergo induction chemotherapy with (TP) docetaxel (Taxotere) 75 mg/m2 and cisplatin 100 mg/m2 (or Carboplatin AUC 6).
  Day #23 (+/- 3 days): Patients will undergo a direct laryngoscopy (DL) with biopsy. Patients will also undergo a repeat CT scan of the neck with perfusion within a week (+/-) of their perspective biopsies.
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: AT-101 — Patients will receive AT-101 40 mg orally two times a day.
  Other Names: Bcl-xL INHIBITOR
  Arms: platinum/docetaxel + AT-101
Drug: Docetaxel — Docetaxel (Taxotere) 75 mg/m2
  Other Names: Taxotere
  Arms: Active Comparator arm
Drug: Cisplatin — Cisplatin 100 mg/m2
Drug: Carboplatin — Carboplatin AUC (area under the curve) 6. Maximum dose of 700 mg

SUMMARY:
To evaluate a new treatment approach for adults with advanced laryngeal cancer: induction chemotherapy with platinum and docetaxel plus AT-101. AT-101 is an investigational drug for the treatment of advanced cancer. It is hoped that the combination of this chemotherapy regimen will allow cancer patients to keep their voice box and to improve/maintain voice-related quality of life. The ultimate goal of this study is to prevent the surgery to remove subjects voice box.

DETAILED DESCRIPTION:
Published data demonstrate equal efficacy and improved quality of life when platinum and a taxane were compared with platinum and 5-Fluorouracil [31]. Additionally, weekly cisplatin regimens (30-40 mg/m2) with radiotherapy appear to be equally efficacious and better tolerated than standard high-dose cisplatin (100 mg/ m2) regimens with radiation therapy for locally advanced SCCHN [32] The investigators will thus attempt to reduce toxicity from induction chemotherapy with the use of docetaxel/cisplatin (or carboplatin) (TP) in place of our previously used standard regimen of cisplatin and 5-fluorouracil (PF) and administer weekly cisplatin (or carboplatin) with radiation for those patients who are responders to induction therapy. Finally, Phase I/II testing of the small molecule inhibitor, AT-101, has recently been completed, and suggests activity in solid tumors when combined with cytotoxic agents. Since the investigators have achieved such high survival rates with our treatment selection approach in laryngeal cancer, our ultimate goal is to reduce the rate of salvage laryngectomy which should improve quality of life. The investigators hypothesize that specific inhibition of Bcl-2/Bcl-xL function can increase response rates to neoadjuvant chemotherapy and decrease the need for salvage laryngectomy. Hence, the investigators propose this study: the treatment of patients with advanced SCC of the larynx with one cycle of platinum plus docetaxel with AT-101, followed by chemoradiotherapy for those responding to this induction regimen and reserving total laryngectomy for those who are non-responders.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed, previously untreated, resectable, squamous cell carcinoma of the larynx or hypopharynx.
* Disease must be Stage III or IV
* Tumor must be potentially surgically resectable and curable with conventional surgery and radiation therapy
* Patients must undergo pre-treatment endoscopic tumor staging and CT scanning
* ECOG Performance status 0-1
* Adequate WBC (white blood cell), granulocyte and platelet counts
* Creatinine clearance of ≥ 60cc/min for cisplatin candidates and ≥ 30 cc/min for carboplatin candidates
* Adequate bilirubin, AST (aspartate aminotransferase), and ALT (alanine transaminase) function

Exclusion Criteria:

* Prior head and neck malignancy or history of other prior non-head and neck malignancy within the past 3 years
* Prior head and neck radiation or prior chemotherapy.
* Documented evidence of distant metastases
* Active infection
* Pregnancy or lactation
* Any medical or psychiatric illness which in the opinion of the principal investigator would compromise the patient's ability to tolerate this treatment
* Patients residing in prison
* Patients with psychiatric/ social situations that would limit compliance with study requirements
* Patients with Grade > 2 peripheral neuropathy
* History of severe hypersensitivity reaction to docetaxel
* Class 3 or 4 cardiac disease
* Unstable angina or history of myocardial ischemia within prior 6 months
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, ulcerative colitis, inflammatory bowel disease, partial or complete small bowel obstruction
* Prior use of gossypol or AT-101, or known hypersensitivity to gossypol or AT-101
* Patients taking any other concurrent approved or investigational anti-cancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2021-11-06 (Actual); Study Completion 2021-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Swiecicki, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: one subject was enrolled; however, disease progression was discovered before active treatment and therefore the patient never was treated with study drug
Groups:
- Platinum/Docetaxal + AT-101: platinum/docetaxel + AT-101 The platinum will either be cisplatin or carboplatin as deemed best by the medical oncologist.
  (Both Arms) Day #1: Patients will undergo induction chemotherapy with (TP) docetaxel (Taxotere) 75 mg/m2 and cisplatin 100 mg/m2 (or Carboplatin AUC 6).
  (AT-101 Arm) Days #1-3: Patients will receive AT-101 40 mg orally twice daily On Day 23 (+/- 3 days), there will be a direct laryngoscopy (DL) with tumor biopsy and blood draw, repeat CT scan of the neck with perfusion within a week biopsy.
  AT-101: Patients will receive AT-101 40 mg orally two times a day.
  Cisplatin: Cisplatin 100 mg/m2
  Carboplatin: Carboplatin AUC (area under the curve) 6. Maximum dose of 700 mg
- Active Comparator Arm: (Both Arms) Day #1: Patients will undergo induction chemotherapy with (TP) docetaxel (Taxotere) 75 mg/m2 and cisplatin 100 mg/m2 (or Carboplatin AUC 6).
  Day #23 (+/- 3 days): Patients will undergo a direct laryngoscopy (DL) with biopsy. Patients will also undergo a repeat CT scan of the neck with perfusion within a week (+/-) of their perspective biopsies.
  Docetaxel: Docetaxel (Taxotere) 75 mg/m2
  Cisplatin: Cisplatin 100 mg/m2
  Carboplatin: Carboplatin AUC (area under the curve) 6. Maximum dose of 700 mg
Period: Overall Study
Arm/Group | Platinum/Docetaxal + AT-101 | Active Comparator Arm
Started | 36 | 18
Completed | 35 | 18
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Platinum/Docetaxal + AT-101: platinum/docetaxel + AT-101 The platinum will either be cisplatin or carboplatin as deemed best by the medical oncologist.
  (Both Arms) Day #1: Patients will undergo induction chemotherapy with (TP) docetaxel (Taxotere) 75 mg/m2 and cisplatin 100 mg/m2 (or Carboplatin AUC 6).
  (AT-101 Arm) Days #1-3: Patients will receive AT-101 40 mg orally twice daily On Day 23 (+/- 3 days), there will be a direct laryngoscopy (DL) with tumor biopsy and blood draw, repeat CT scan of the neck with perfusion within a week biopsy.
  AT-101: Patients will receive AT-101 40 mg orally two times a day.
  Cisplatin: Cisplatin 100 mg/m2
  Carboplatin: Carboplatin AUC (area under the curve) 6. Maximum dose of 700 mg
  Per physician discretion, carboplatin was used in lieu of cisplatin for 13 patients in this arm
- Active Comparator Arm: (Both Arms) Day #1: Patients will undergo induction chemotherapy with (TP) docetaxel (Taxotere) 75 mg/m2 and cisplatin 100 mg/m2 (or Carboplatin AUC 6).
  Day #23 (+/- 3 days): Patients will undergo a direct laryngoscopy (DL) with biopsy. Patients will also undergo a repeat CT scan of the neck with perfusion within a week (+/-) of their perspective biopsies.
  Docetaxel: Docetaxel (Taxotere) 75 mg/m2
  Cisplatin: Cisplatin 100 mg/m2
  Per physician discretion, carboplatin was used in lieu of cisplatin for 10 patients in this arm Carboplatin: Carboplatin AUC (area under the curve) 6. Maximum dose of 700 mg
- Total: Total of all reporting groups
Arm/Group | Platinum/Docetaxal + AT-101 | Active Comparator Arm | Total
Number analyzed (Participants) | 36 | 18 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 11 | 38
  >=65 years | 9 | 7 | 16
Age, Continuous [Mean (Full Range); unit: years] | 58.5 [19 to 82] | 61.4 [33 to 77] | 59.95 [19 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 0 | 8
  Male | 28 | 18 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 35 | 18 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 18 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Alive and Free From Indication for Laryngectomy Three Months Post Treatment
Description: The primary clinical objective of this trial is to compare the larynx preservation rates in a treatment paradigm that uses induction chemotherapy plus AT-101 to select patients for either concurrent chemoradiation or surgery. Organ preservation rate, defined as alive and free from indication for laryngectomy three months post treatment, was chosen as the primary endpoint because it provides evidence to fully characterize clinically the effect of the treatment strategy
Time Frame: Up to 3 months after end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum/Docetaxal + AT-101 | Active Comparator Arm
Number analyzed (Participants) | 34 | 18
Participants | 27 | 12

2. Primary Outcome: Progression-free Survival
Description: Time from randomization to the time of first indication of local failure or metastases. Estimated non-parametrically using the Kaplan-Meier method.
Time Frame: Up to 3 years after randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Platinum/Docetaxal + AT-101: platinum/docetaxel + AT-101 The platinum will either be cisplatin or carboplatin as deemed best by the medical oncologist.
  Patients underwent induction chemotherapy with (TP) docetaxel (Taxotere) 75 mg/m2 and cisplatin 100 mg/m2 (or Carboplatin AUC 6).
  (AT-101 Arm) Days #1-3: Patients received AT-101 40 mg orally twice daily On Day 23 (+/- 3 days), there will be a direct laryngoscopy (DL) with tumor biopsy and blood draw, repeat CT scan of the neck with perfusion within a week biopsy.
  AT-101: Patients received AT-101 40 mg orally two times a day.
  Cisplatin: Cisplatin 100 mg/m2
  Carboplatin: Carboplatin AUC (area under the curve) 6. Maximum dose of 700 mg
- Active Comparator Arm: Patients underwent induction chemotherapy with (TP) docetaxel (Taxotere) 75 mg/m2 and cisplatin 100 mg/m2 (or Carboplatin AUC 6).
  Day #23 (+/- 3 days): Patients underwent a direct laryngoscopy (DL) with biopsy. Patients also underwent a repeat CT scan of the neck with perfusion within a week (+/-) of their perspective biopsies.
  Docetaxel: Docetaxel (Taxotere) 75 mg/m2
  Cisplatin: Cisplatin 100 mg/m2
  Carboplatin: Carboplatin AUC (area under the curve) 6. Maximum dose of 700 mg
Arm/Group | Platinum/Docetaxal + AT-101 | Active Comparator Arm
Number analyzed (Participants) | 31 | 15
percentage of participants | 55 [35 to 71] | 65 [36 to 84]

3. Primary Outcome: Overall Response Rate (ORR)
Description: ORR (Complete Response [CR] plus Partial Response [PR]) to induction chemotherapy with platinum and docetaxel plus AT-101 following one and/or two cycles in patients with advanced laryngeal cancer.
Time Frame: Up to approximately 60 days
Population: This outcome measure only applies to those subjects treated with induction chemotherapy with platinum and docetaxel plus AT-101 and therefore only one arm is being reported
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum/Docetaxal + AT-101
Number analyzed (Participants) | 36
Participants | 27

4. Primary Outcome: Percentage of Patients Experiencing Grade 3 or Higher Adverse Events.
Description: Toxicities will be evaluated using the Common Terminology Criteria for Adverse Events (CTCAE), version 3.
Time Frame: Up to 3 years after end of treatment
Measure: Number; unit: percentage of Patients
Arm/Group | Platinum/Docetaxal + AT-101 | Active Comparator Arm
Number analyzed (Participants) | 36 | 18
percentage of Patients | 61 | 44

5. Secondary Outcome: Head and Neck Related Quality of Life (QOL)
Description: University of Michigan Head and Neck Quality of Life Instrument (HN-QOL) will be administered prior to treatment (i.e. pre-induction chemotherapy) and at 6 months, 12 months, and 24 months (+/- 4 months) after completion of chemo-RT or surgery-RT (or surgery-chemoRT, as indicated). Scale is 0-100 with high scores indicating a better outcome.
Time Frame: Up to 28 months post treatment
Population: Number of participants analyzed varies below based on completion compliance
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Platinum/Docetaxal + AT-101 | Active Comparator Arm
Number analyzed (Participants) | 36 | 18
units on a scale
  Emotion- Prior to treatment: number analyzed (Participants) | 35 | 17
  Emotion- Prior to treatment | 66.7 [41.7 to 79.2] | 62.5 [58.3 to 75]
  Emotion- 6 months: number analyzed (Participants) | 24 | 11
  Emotion- 6 months | 66.7 [41.7 to 95.8] | 95.8 [75.0 to 100]
  Emotion- 12 months: number analyzed (Participants) | 22 | 11
  Emotion- 12 months | 72.9 [66.7 to 83.3] | 91.7 [75 to 100]
  Emotion- 24 months: number analyzed (Participants) | 16 | 9
  Emotion- 24 months | 75 [52.1 to 81.3] | 91.7 [91.7 to 95.8]
  Speech- Prior to treatment | 46.9 [37.5 to 62.5] | 34.4 [25 to 68.8]
  Speech- 6 Months: number analyzed (Participants) | 24 | 11
  Speech- 6 Months | 56.3 [21.9 to 78.1] | 50 [37.5 to 81.3]
  Speech- 12 Months: number analyzed (Participants) | 23 | 11
  Speech- 12 Months | 50 [31.3 to 75] | 62.5 [18.8 to 87.5]
  Speech- 24 Months: number analyzed (Participants) | 15 | 9
  Speech- 24 Months | 50 [43.8 to 75] | 75 [50 to 87.5]
  Pain- Prior to treatment: number analyzed (Participants) | 36 | 17
  Pain- Prior to treatment | 59.4 [43.8 to 75] | 68.8 [56.3 to 87.5]
  Pain- 6 months: number analyzed (Participants) | 24 | 11
  Pain- 6 months | 62.5 [31.3 to 87.5] | 81.3 [62.5 to 87.5]
  Pain- 12 months: number analyzed (Participants) | 23 | 10
  Pain- 12 months | 68.8 [43.8 to 91.7] | 62.5 [58.3 to 87.5]
  Pain- 24 months: number analyzed (Participants) | 16 | 9
  Pain- 24 months | 56.3 [28.1 to 87.5] | 87.5 [75 to 93.8]

6. Secondary Outcome: Voice Related QOL
Description: The University of Michigan Voice Related Quality of Life Measure (V-RQOL) will be administered prior to treatment (i.e. pre-induction chemotherapy) and at 6 months, 12 months, and 24 months (+/- 4 months) after completion of chemo-RT or surgery-RT (or surgery-chemoRT, as indicated). Scale is 0-50 (10 items scale 1-5) with high scores indicating a worse outcome.
Time Frame: Up to 28 months post treatment
Population: number of participants analyzed varies due to patient compliance and patients coming off trial per protocol
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Platinum/Docetaxal + AT-101 | Active Comparator Arm
Number analyzed (Participants) | 35 | 17
score on a scale
  VRQOL-SUM- Prior to treatment | 25 [18 to 29] | 24 [20 to 34]
  VRQOL-SUM- 6 Months: number analyzed (Participants) | 22 | 11
  VRQOL-SUM- 6 Months | 23 [13 to 32] | 23 [14 to 28]
  VRQOL-SUM- 12 Months: number analyzed (Participants) | 20 | 9
  VRQOL-SUM- 12 Months | 26 [17 to 32.5] | 22 [13 to 31]
  VRQOL-SUM- 24 Months: number analyzed (Participants) | 13 | 9
  VRQOL-SUM- 24 Months | 22 [15 to 32] | 21 [15 to 23]
  NOISY_VAL_- Prior to treatment | 4 [3 to 4] | 4 [3 to 4]
  NOISY_VAL_- 6months: number analyzed (Participants) | 22 | 11
  NOISY_VAL_- 6months | 3 [2 to 4] | 3 [2 to 5]
  NOISY_VAL_- 12 months: number analyzed (Participants) | 20 | 9
  NOISY_VAL_- 12 months | 4 [3 to 4.5] | 3 [2 to 4]
  NOISY_VAL_- 24 months: number analyzed (Participants) | 13 | 9
  NOISY_VAL_- 24 months | 3 [2 to 5] | 4 [3 to 4]
  OUTOFAIR_VAL- Prior to treatment | 2 [1 to 2] | 2 [1 to 3]
  OUTOFAIR_VAL- 6 months: number analyzed (Participants) | 22 | 11
  OUTOFAIR_VAL- 6 months | 2 [1 to 3] | 1 [1 to 3]
  OUTOFAIR_VAL- 12 months: number analyzed (Participants) | 20 | 9
  OUTOFAIR_VAL- 12 months | 2 [1 to 3] | 2 [1 to 3]
  OUTOFAIR_VAL- 24 months: number analyzed (Participants) | 13 | 9
  OUTOFAIR_VAL- 24 months | 2 [1 to 3] | 1 [1 to 3]
  WHATCOMEOUT_VAL_3n- Prior to treatment | 1 [1 to 3] | 1 [1 to 3]
  WHATCOMEOUT_VAL_3n- 6 months: number analyzed (Participants) | 22 | 11
  WHATCOMEOUT_VAL_3n- 6 months | 2 [1 to 3] | 2 [1 to 3]
  WHATCOMEOUT_VAL_3n- 12 months: number analyzed (Participants) | 20 | 9
  WHATCOMEOUT_VAL_3n- 12 months | 2 [1 to 2] | 1 [1 to 3]
  WHATCOMEOUT_VAL_3n- 24 months: number analyzed (Participants) | 13 | 9
  WHATCOMEOUT_VAL_3n- 24 months | 2 [1 to 3] | 2 [1 to 2]
  ANXIOUS_VAL_4n- Prior to treatment | 3 [1 to 4] | 3 [2 to 3]
  ANXIOUS_VAL_4n- 6 months: number analyzed (Participants) | 22 | 11
  ANXIOUS_VAL_4n- 6 months | 3 [1 to 4] | 2 [1 to 3]
  ANXIOUS_VAL_4n- 12 months: number analyzed (Participants) | 20 | 9
  ANXIOUS_VAL_4n- 12 months | 2.5 [2 to 4] | 2 [1 to 3]
  ANXIOUS_VAL_4n- 24 months: number analyzed (Participants) | 13 | 9
  ANXIOUS_VAL_4n- 24 months | 3 [2 to 4] | 2 [1 to 4]
  DEPRESSED_VAL_5n- Prior to treatment | 2 [1 to 3] | 2 [1 to 3]
  DEPRESSED_VAL_5n- 6 months: number analyzed (Participants) | 22 | 11
  DEPRESSED_VAL_5n- 6 months | 2 [1 to 3] | 1 [1 to 2]
  DEPRESSED_VAL_5n- 12 months: number analyzed (Participants) | 20 | 9
  DEPRESSED_VAL_5n- 12 months | 2 [1 to 3] | 1 [1 to 1]
  DEPRESSED_VAL_5n- 24 months: number analyzed (Participants) | 13 | 9
  DEPRESSED_VAL_5n- 24 months | 2 [1 to 4] | 1 [1 to 2]
  TROUBLEPHONE_VAL_6n- Prior to treatment | 3 [2 to 4] | 3 [3 to 4]
  TROUBLEPHONE_VAL_6n- 6 Months: number analyzed (Participants) | 22 | 11
  TROUBLEPHONE_VAL_6n- 6 Months | 2 [2 to 4] | 2 [1 to 4]
  TROUBLEPHONE_VAL_6n- 12 Months: number analyzed (Participants) | 20 | 9
  TROUBLEPHONE_VAL_6n- 12 Months | 3 [2 to 4] | 3 [1 to 3]
  TROUBLEPHONE_VAL_6n- 24 Months: number analyzed (Participants) | 13 | 9
  TROUBLEPHONE_VAL_6n- 24 Months | 3 [1 to 4] | 2 [2 to 2]
  TROUBLEJOB_VAL_7n- Prior to treatment | 2 [1 to 3] | 2 [1 to 4]
  TROUBLEJOB_VAL_7n- 6 Months: number analyzed (Participants) | 22 | 11
  TROUBLEJOB_VAL_7n- 6 Months | 1 [1 to 4] | 1 [1 to 2]
  TROUBLEJOB_VAL_7n- 12 Months: number analyzed (Participants) | 20 | 9
  TROUBLEJOB_VAL_7n- 12 Months | 2.5 [1 to 3] | 1 [1 to 3]
  TROUBLEJOB_VAL_7n- 24 Months: number analyzed (Participants) | 13 | 9
  TROUBLEJOB_VAL_7n- 24 Months | 2 [1 to 4] | 1 [1 to 2]
  AVOIDSOCIALLY_VAL_8n- Prior to treatment | 1 [1 to 2] | 2 [1 to 4]
  AVOIDSOCIALLY_VAL_8n- 6 months: number analyzed (Participants) | 22 | 11
  AVOIDSOCIALLY_VAL_8n- 6 months | 2 [1 to 3] | 2 [1 to 4]
  AVOIDSOCIALLY_VAL_8n- 12 months: number analyzed (Participants) | 20 | 9
  AVOIDSOCIALLY_VAL_8n- 12 months | 1.5 [1 to 3] | 2 [1 to 3]
  AVOIDSOCIALLY_VAL_8n- 24 months: number analyzed (Participants) | 13 | 9
  AVOIDSOCIALLY_VAL_8n- 24 months | 2 [1 to 3] | 1 [1 to 2]
  REPEATMYSELF_VAL_9n- Prior to treatment | 3 [2 to 4] | 3 [2 to 4]
  REPEATMYSELF_VAL_9n- 6 months: number analyzed (Participants) | 22 | 11
  REPEATMYSELF_VAL_9n- 6 months | 3 [2 to 4] | 3 [2 to 4]
  REPEATMYSELF_VAL_9n- 12 months: number analyzed (Participants) | 20 | 9
  REPEATMYSELF_VAL_9n- 12 months | 3 [2 to 4] | 3 [2 to 4]
  REPEATMYSELF_VAL_9n- 24 months: number analyzed (Participants) | 13 | 9
  REPEATMYSELF_VAL_9n- 24 months | 2 [1 to 4] | 3 [2 to 4]
  LESSOUTGOING_VAL_10n- Prior to treatment | 2 [1 to 3] | 3 [1 to 4]
  LESSOUTGOING_VAL_10n- 6 months: number analyzed (Participants) | 22 | 11
  LESSOUTGOING_VAL_10n- 6 months | 2 [1 to 4] | 2 [1 to 3]
  LESSOUTGOING_VAL_10n- 12 months: number analyzed (Participants) | 20 | 9
  LESSOUTGOING_VAL_10n- 12 months | 2 [1 to 3] | 2 [1 to 3]
  LESSOUTGOING_VAL_10n- 24 months: number analyzed (Participants) | 13 | 9
  LESSOUTGOING_VAL_10n- 24 months | 2 [1 to 3] | 2 [1 to 2]

7. Secondary Outcome: Functional Assessment QOL
Description: University of Michigan Head and Neck Quality of Life Instrument (HN-QOL) will be administered prior to treatment (i.e. pre-induction chemotherapy) and at 6 months, 12 months, and 24 months (+/- 4 months) after completion of chemo-RT or surgery-RT (or surgery-chemoRT, as indicated). Scale is 0-100 with high scores indicating a better outcome. EATING Domain is reported here as a functional assessment.
Time Frame: Up to 28 months post treatment
Population: Number of participants analyzed varies below based on completion compliance
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Platinum/Docetaxal + AT-101 | Active Comparator Arm
Number analyzed (Participants) | 36 | 18
score on a scale
  EATING- Prior to treatment: number analyzed (Participants) | 36 | 11
  EATING- Prior to treatment | 83.3 [64.6 to 93.8] | 91.7 [83.3 to 100]
  EATING- 6 months: number analyzed (Participants) | 24 | 18
  EATING- 6 months | 75 [60.4 to 85.4] | 83.3 [75 to 87.5]
  EATING- 12 months: number analyzed (Participants) | 23 | 9
  EATING- 12 months | 83.3 [66.7 to 91.7] | 83.3 [62.5 to 87.5]
  EATING- 24 months: number analyzed (Participants) | 16 | 9
  EATING- 24 months | 77.1 [67.7 to 87.5] | 95.8 [75 to 95.8]

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 30 days after the last dose of study treatment; additionally, any serious adverse event occurring more than 30 days after the last study treatment if considered to be related to the study treatment. Data was collected during a 6.5 year period.
Arm/Group | Platinum/Docetaxal + AT-101 | Active Comparator Arm
All-Cause Mortality (participants affected / at risk) | 1/36 | 1/18
Serious Adverse Events (participants affected / at risk) | 14/36 | 5/18
Other Adverse Events (participants affected / at risk) | 36/36 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Platinum/Docetaxal + AT-101 (N=36) | Active Comparator Arm (N=18)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic reaction (General disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Disease Progression (General disorders) | 0 (0) | 1 (1) — Cause of death larynx cancer.
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Squamous Cell Carcinoma - Nose (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1)
Acute Kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperkalemia (Investigations) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypokalemia (Investigations) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infection, Lung (pneumonia) (Infections and infestations) | 0 (0) | 2 (2)
Infection, Upper aerodigestive NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection, Upper airway NOS (Infections and infestations) | 1 (1) | 0 (0)
Intracranial hemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neck pain (General disorders) | 1 (1) | 0 (0)
neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (3) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
pulmonary embolism (Cardiac disorders) | 1 (1) | 0 (0)
Tracheal hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Platinum/Docetaxal + AT-101 (N=36) | Active Comparator Arm (N=18)
Abdominal distention (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acne (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2) | 3 (5)
Allergic reaction (Immune system disorders) | 2 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 7 (7) | 5 (6)
Anxiety (Psychiatric disorders) | 9 (9) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (7) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 10 (11) | 9 (10)
Constitutional Symptoms - Other (Specify) (General disorders) | 1 (1) | 0 (0) — BUN Increase
Constitutional Symptoms - Other (Specify) (General disorders) | 0 (0) | 1 (1) — restless leg syndrome
Constitutional Symptoms - Other (Specify) (General disorders) | 1 (1) | 0 (0) — paronychia of left thumb
Constitutional Symptoms - Other (Specify) (General disorders) | 1 (1) | 0 (0) — increase mucus in throat
Constitutional Symptoms - Other (Specify) (General disorders) | 0 (0) | 1 (1) — orthostatic
cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
Creatinine increased (Investigations) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 3 (3)
Dermal change (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis radiation (Skin and subcutaneous tissue disorders) | 7 (9) | 3 (3)
Dermatology/Skin - Other (Specify) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — skin changes
Dermatology/Skin - Other (Specify) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — cut on the right hand
Dermatology/Skin - Other (Specify) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — psoriasis flare up on lower right and left arms
Dermatology/Skin - Other (Specify) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — psoriasis flare up on abdomen
Dermatology/Skin - Other (Specify) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — drainage from neck incisions
Dermatology/Skin - Other (Specify) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — hydration infusion site swelling
Diarrhea (Gastrointestinal disorders) | 16 (16) | 6 (7)
Dizziness (Nervous system disorders) | 7 (7) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 16 (18) | 6 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 15 (23) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear, nose and throat examination abnormal (Ear and labyrinth disorders) | 7 (8) | 2 (2)
Edema limbs (General disorders) | 6 (8) | 1 (1)
Edema: head and neck (General disorders) | 3 (3) | 0 (0)
Edema: viscera (General disorders) | 2 (3) | 2 (3)
Erythema multiforme (General disorders) | 1 (1) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 2 (3) | 3 (5)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 8 (14) | 3 (4)
External ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 15 (16) | 10 (13)
Fever (General disorders) | 3 (3) | 0 (0)
Flu-like syndrome (General disorders) | 0 (0) | 1 (1)
Fracture (General disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI - Other (Specify) (Gastrointestinal disorders) | 0 (0) | 1 (1) — hametochezia
GI - Other (Specify) (Gastrointestinal disorders) | 1 (1) | 0 (0) — indigestion
GI - Other (Specify) (Gastrointestinal disorders) | 0 (0) | 1 (1) — increase reflux symptoms
Hand-and-foot syndrome (General disorders) | 2 (2) | 2 (3)
Headache (General disorders) | 4 (5) | 0 (0)
Hearing (without monitoring program) (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Heartburn (General disorders) | 0 (0) | 1 (1)
Hemoglobin decrease (Investigations) | 6 (11) | 6 (10)
Hemorrhage - Other (Specify) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — hemoptysis
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hyperbilirubinemia (Investigations) | 1 (1) | 0 (0)
Hypercalcemia (Investigations) | 2 (3) | 0 (0)
Hyperglycemia (Investigations) | 4 (17) | 1 (3)
Hyperkalemia (Investigations) | 2 (2) | 1 (2)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Investigations) | 2 (4) | 1 (1)
Hypocalcemia (Investigations) | 4 (7) | 1 (1)
Hypokalemia (Investigations) | 3 (4) | 0 (0)
Hypomagnesemia (Investigations) | 3 (3) | 0 (0)
Hyponatremia (Investigations) | 4 (7) | 2 (4)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Infection - Other (Specify) (Infections and infestations) | 1 (1) | 0 (0) — thrush
Infection - Other (Specify) (Infections and infestations) | 1 (1) | 0 (0) — pneumonia
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0)
Intraoperative ocular injury (Eye disorders) | 1 (1) | 0 (0)
Involuntary movement (Nervous system disorders) | 0 (0) | 1 (1)
Joint pain (General disorders) | 1 (1) | 1 (1)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Laryngoscopy abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 8 (9) | 7 (7)
Mucositis oral (Gastrointestinal disorders) | 5 (5) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal - Other (Specify) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — muscle twitching
Musculoskeletal - Other (Specify) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — DHT discomfort
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 23 (43) | 11 (15)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
neutropenia (Investigations) | 5 (6) | 3 (3)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 7 (9) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (6) | 3 (3)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 7 (8)
Platelet count decreased (Investigations) | 10 (15) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Radiation recall reaction (dermatologic) (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 8 (11) | 4 (5)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
chills (General disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Vascular disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Taste alteration (Nervous system disorders) | 21 (25) | 6 (11)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 8 (9) | 5 (5)
Toothache (General disorders) | 1 (1) | 1 (1)
Tracheostomy site bleeding (General disorders) | 0 (0) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Tumor pain (General disorders) | 2 (2) | 0 (0)
Upper aerodigestive tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Voice alteration (General disorders) | 6 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 13 (19) | 2 (2)
Weight gain (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 12 (18) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT01633541/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT01633541/ICF_001.pdf